CLINICAL TRIAL: NCT01917357
Title: A Phase III, Open-label, Randomized Parallel-group Study on the Immunogenicity and Safety of Quinvaxem® DTwP-HepB-Hib) in Uniject™ With Quinvaxem® Monodose Vials in Healthy Infants at 6, 10 and 14 Weeks of Age
Brief Title: A Comparison of the Immunogenicity and Safety of Quinvaxem in Mono-dose Vials and Uniject
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: QVX-V-D001
Record Dates: First submitted 2013-08-05; First posted 2013-08-06 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-02

CONDITIONS: Diphtheria; Pertussis; Tetanus; Hepatitis B; Haemophilus Infections
Keywords: Vaccination; Immunisation; Virus; Diphtheria; Pertussis; Tetanus; Hepatitis B; Haemophilus Influenzae; Immunity
MeSH Terms: conditions — Diphtheria; Whooping Cough; Tetanus; Hepatitis B; Haemophilus Infections; Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quinvaxem in Uniject (Experimental): A single dose (0.5 mL) of Quinvaxem contains:
  diphtheria antitoxin (>= 30 IU), tetanus antitoxin (>= 60 IU), whole-cell inactive pertussis bacteria (>= 4 IU), 10 mcg Hib oligosaccharide conjugate (approx. 25 mcg CRM197), 10 mcg Hepatitis B surface antigen
  One dose of Quinvaxem given intramuscularly at Weeks 6, 10 and 14 by injection into the anterolateral region of the thigh using the Uniject pre-filled injection device
  Interventions: Biological: Quinvaxem in Uniject
- Quinvaxem in single dose vials (Active Comparator): A single dose (0.5 mL) of Quinvaxem contains:
  diphtheria antitoxin (>= 30 IU), tetanus antitoxin (>= 60 IU), whole-cell inactive pertussis bacteria (>= 4 IU), 10 mcg Hib oligosaccharide conjugate (approx. 25 mcg CRM197), 10 mcg Hepatitis B surface antigen
  One dose of Quinvaxem given intramuscularly at Weeks 6, 10 and 14 by injection into the anterolateral region of the thigh using a needle and syringe from single dose vials
  Interventions: Biological: Quinvaxem in single dose vials

INTERVENTIONS:
Biological: Quinvaxem in Uniject
  Arms: Quinvaxem in Uniject
Biological: Quinvaxem in single dose vials
  Arms: Quinvaxem in single dose vials

SUMMARY:
This is a study to show that vaccination with three doses of Quinvaxem presented in Uniject is not inferior to vaccination with three doses of Quinvaxem presented in single dose vials, with respect to protection against all antibodies (anti-hepatitis B surface antibodies, anti-polyribosyl ribitol phosphate (PRP), anti-diphtheria, anti-tetanus and anti-Bordetella pertussis) one (1) month after completion of the 6-10-14 week vaccination course.

ELIGIBILITY:
Inclusion Criteria:

* A male or female between, and including, 42 and 64 days of age at the time of the first vaccination
* Written informed consent obtained from parents/legal guardians of the subject
* Free of obvious health problems as established by medical history and/or clinical examination before entering the study
* HepB vaccination at birth (within 48 hours)
* Available for all scheduled study visits

Exclusion Criteria:

* Use of any investigational drug or any investigational vaccine in the 30 days preceding the first dose of study vaccine, or their planned use during the study period and safety follow-up
* Planned administration of a vaccine not foreseen by the Study Protocol
* Known or suspected impairment of immune function, known HIV-positivity; actively receiving immunosuppressive therapy, or in receipt of systemic immunosuppressive therapy in the one month prior to study entry (note: inhaled and topical steroids are allowed)
* Administration of parenteral immunoglobulin preparation and/or blood products since birth
* Previous vaccination against Hib and/or DTP
* History of anaphylaxis, or any serious vaccine reaction, or hypersensitivity to any vaccine component or to products containing mercury compounds, such as thiomersal
* Clinically significant acute infection
* Clinically significant acute illness
* Any condition that, in the opinion of the investigator, might interfere with the evaluation of the study objectives
* Participation in another clinical study

Ages: 42 Days to 64 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2013-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Seroprotection Rate: Anti-PRP Antibodies | 1 month after the third vaccination
Seroprotection Rate: Anti-hepatitis B Surface Antibodies | 1 month after the third vaccination
Anti-diphtheria Toxoid Antibodies | 1 month after the third vaccination
Seroprotection Rate: Anti-tetanus Toxoid Antibodies | 1 month after the third vaccination
Seroprotection Rate: Anti-B. Pertussis Antibodies | 1 month after the third vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Maria RZ Capeding, MD, Principal Investigator — Research Institute for Tropical Medicine (RITM)
Locations (1):
- Research Institute for Tropical Medicine, City of Muntinlupa, Philippines